CLINICAL TRIAL: NCT02606591
Title: Houston Independent School District (HISD) Yoga and Wellness Program Evaluation
Brief Title: Houston Independent School District (HISD) Yoga Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PA15-0677
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Health and Wellness
Keywords: Electroencephalograph; EEG; Hair sample; Cognitive tests; Cortisol analysis; Brain activity; Stress hormones
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroencephalograph (EEG) + Testing (Experimental): Participants complete an electroencephalograph (EEG) cognitive tests, and provide a hair sample shortly after entering the study and again near the end of the school year. Hair sample tested to measure a stress hormone called cortisol.
  Interventions: Procedure: Electroencephalograph; Behavioral: Cognitive Tests; Other: Hair Sample

INTERVENTIONS:
Procedure: Electroencephalograph — EEG performed at beginning and end of school year.
  Other Names: EEG
Behavioral: Cognitive Tests — During the EEG, participant asked to wear headphones and do some simple tests on the computer that measure their abilities to see, hear, and understand information.
Other: Hair Sample — Participants provide a sample of hair at baseline (near the beginning of school), and follow-up (near the end of school). Sample tested to measure cortisol levels.

SUMMARY:
The goal of this research study is to learn about how brain activity, cognitive tests (tests of participant's brain function), and stress hormones are related to taking part in a health and wellness program in elementary-aged students.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, they will complete an electroencephalograph (EEG -- a test that measures the electrical activity of the brain), cognitive tests, and provide a hair sample shortly after they enter the study and again near the end of the school year.

The testing will take place in a room at participant's school chosen by the teachers. A member of the study staff will walk participant from their classroom and be with them the whole time the testing is taking place and then take them back to their classroom. If the testing is done before or after school, participant will stay with the member of study staff until their parent or guardian comes to pick them up.

During the EEG, researchers will place 19 electrodes on participant's head and 1 or 2 electrodes on each earlobe. Gel will be used to help attach the electrodes. The electrodes will measure and record participant's brain wave activity, similar to the way a doctor listens to their heart beat from the surface of their skin. During the EEG, participant will be also asked to wear headphones and do some simple tests on the computer that measure their abilities to see, hear, and understand information. The EEG will take up to 5 minutes to set up and then 25 minutes for testing.

Participant will also provide a sample of hair, about 75 strands which is like the thickness of a pencil. The hair will tested to measure a stress hormone called cortisol. The hair will be destroyed after study testing.

Data obtained from the hair samples and EEG will be analyzed alongside the data participant is providing our collaborators at the University of San Diego and the Houston Independent School District.

The EEG that is collected for this study is for research purposes only. It is not the same as a "clinical EEG" that is used in medical diagnosis. The EEG that the study staff will collect looks at how the brain functions. It is not designed to look for medical conditions, the way that an MRI or CAT scan would be used. However, if a possible medical condition is suspected, participant will be told to follow up with their medical provider.

Length of Participation:

Participation on this study will be over after participant provides a hair sample, complete the EEG, and complete the cognitive tests the second time near the end of the school year.

This is an investigational study.

Up to 200 participants will be enrolled in this study. All will take part through MD Anderson at their schools.

ELIGIBILITY:
Inclusion Criteria:

1. Fourth and Fifth graders in Houston Independent School District (HISD) schools that are participating in the Sonima Foundation's Health and Wellness Program
2. Participant on USD study protocol.

Exclusion Criteria: 1)

1. Participants who are taking any antipsychotic medications
2. Participants with active central nervous system (CNS) disease or encephalopathy
3. Participants who have ever been diagnosed with bipolar disorder or schizophrenia
4. Participants who have a history of head injury or who have a known seizure activity.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of Collecting Electroencephalograms (EEGs; for Brain Activity Analysis in Elementary-Aged Children Participating in a Health and Wellness Program | 9 months
  Trial feasible if 50% of students who are enrolled complete the EEG's.
Feasibility of Collecting Hair Samples (for Cortisol Analysis) in Elementary-Aged Children Participating in a Health and Wellness Program | 9 months
  Trial feasible if 50% of students who are enrolled submit hair samples.

SECONDARY OUTCOMES:
Changes in EEG During Each State (Eyes Open, Eyes Closed, and During Cognitive Testing) | At baseline and at 9 months
  Changes in EEG during each state (eyes open, eyes closed, and during cognitive testing) assessed using LORETA EEG analysis of brain function at baseline and the follow-up time point acquired through a Mitstar amplifier using WinEEG software.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org